CLINICAL TRIAL: NCT00876889
Title: Safety and Pharmacokinetics of Riluzole in Patients With Traumatic Acute Spinal Cord Injury
Brief Title: Safety of Riluzole in Patients With Acute Spinal Cord Injury
Status: Completed | Type: Observational
Sponsor: The Methodist Hospital Research Institute (Other)
Collaborators: Christopher Reeve Paralysis Foundation (Other); United States Department of Defense (U.S. Federal Agency); AO Clinical Investigation and Publishing Documentation (Other); Ontario Neurotrauma Foundation (Other)
Responsible Party: Principal Investigator, Robert G. Grossman, MD, Professor, Department of Neurosurgery, The Methodist Hospital Research Institute
Other Study IDs: Pro00002029; W81XWH-07-0042 (Other: Department of Defense)
Record Dates: First submitted 2009-03-25; First posted 2009-04-07 (Estimated); Last update posted 2017-09-12 (Actual); Status verified 2017-09

CONDITIONS: Spinal Cord Injury
Keywords: spinal cord injury; riluzole; pharmacokinetics; Acute Traumatic Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Riluzole

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma and cerebral spinal fluid
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Riluzole — 50mg PO (by mouth) every 12 hours starting within 12 hours of injury and continuing for 14 days (28 doses).
  Other Names: Rilutek

SUMMARY:
The purpose of the study is to find out if the use of the drug Riluzole is both safe and improves outcome in patients with acute traumatic spinal cord injury (SCI).

DETAILED DESCRIPTION:
The primary aim of the study is to develop acute care safety and pharmacokinetic profiles of riluzole in patients who have sustained a acute traumatic spinal cord injury. Secondary objectives are to conduct exploratory analyses of functional outcomes for purposes of planning a subsequent Phase II randomized study of the efficiency of Riluzole for the treatment of acute traumatic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

* Age equal to or greater than 18 years and less than or equal to 70 years;
* Willing to give written informed consent to participate in the study. The informed consent may require legally authorized representative to sign if arm/hand function is compromised.
* No other life-threatening injury
* Spinal cord injury at the neurologic level from C4 to T12
* ASIA Impairment Scale level A, B or C
* No cognitive impairment which would preclude an informed consent (including moderate or severe traumatic brain injury)
* Less than 12 hours since injury

Exclusion Criteria:

* Equal or more than 12 hours since injury
* Hypersensitivity to riluzole or any of its components
* Unable to receive riluzole orally or via nasogastric tube
* History of liver or kidney disease (e.g. Hepatitis A, B or C, Cirrhosis, etc.)
* Has a recent history of regular substance abuse (illicit drugs, alcohol)
* Unconscious
* Penetrating spinal cord injury
* Pregnancy as established by urine pregnancy test
* Breastfeeding
* Life expectancy less than 12 months
* Is currently involved in another therapeutic SCI research study that precludes or complicates participation in this study (e.g. study of another therapeutic drug aiming for spinal cord injury recovery, any study that substantially interferes with the follow -up schedule (f/u) schedule, or any high risk study that complicates evaluation of safety outcomes. Types of studies that would not preclude participation are e.g. behavioral adaptation studies, mental health interventions)
* Has a mental disorder or other illness, which in the view of the site investigator, would preclude accurate evaluation (e.g. schizophrenia, severe cognitive disability, Parkinson disease)
* Unable to commit to the follow-up schedule
* Is a prisoner
* Unable to converse, read or write English at the elementary school level

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Admitted to a NACTN hospital
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2010-04; Primary Completion 2011-06 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
American Spinal Injury Association Impairment Scale | Baseline, days 3 and 14, 6 weeks, 3 and 6 months and unscheduled follow-up
  Neurological assessment and classification of spinal cord injury

CONTACTS AND LOCATIONS:
Overall Officials: Robert G Grossman, MD, Study Chair — The Methodist Hospital Research Institute; Michael Fehlings, MD, PhD, Principal Investigator — University of Toronto/Toronto Western Hospital, Toronto; Michele M Johnson, MD, Principal Investigator — the University of Houston/Memorial HermannHospital, Houston; Christopher Shaffery, MD, Principal Investigator — University of Virginia Health System, Charlottesville; Susan Harkema, PhD, Principal Investigator — University of Louisville, Louisville; Bizhan Aarabi, MD, Principal Investigator — University of Maryland Medical Center, Baltimore; James Harrop, MD, Principal Investigator — Thomas Jefferson University, Philadelphia; James Guest, MD, PhD, Principal Investigator — University of Miami, Miami; Ralph Frankowski, PhD, Principal Investigator — The University of Texas School of Public Health, Houston; Diana Chow, PhD, Principal Investigator — University of Houston, College of Pharmacy, Houston
Locations (8):
- United States (7):
  - University of Miami, Miami, Florida
  - University of Louisville Health Sciences Center, Louisville, Kentucky
  - University of Maryland Medical Center, Baltimore, Maryland
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - The Methodist Hospital, Houston, Texas
  - The University of Texas, Houston, Texas
  - University of Virginia Health System, Charlottesville, Virginia
- University of Toronto/Toronto Western Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Carroll AH, Fakhre E, Quinonez A, Tannous O, Mesfin A. An Update on Spinal Cord Injury and Current Management. JBJS Rev. 2024 Oct 24;12(10). doi: 10.2106/JBJS.RVW.24.00124. eCollection 2024 Oct 1. PMID 39446982
- [Derived] Chow DS, Nguyen A, Park J, Wu L, Toups EG, Harrop JS, Guest JD, Schmitt KM, Aarabi B, Fehlings MG, Boakye M, Grossman RG. Riluzole in Spinal Cord Injury Study (RISCIS)-Pharmacokinetic (PK) Sub-Study: An Analysis of Pharmacokinetics, Pharmacodynamics, and Impact on Axonal Degradation of Riluzole in Patients With Traumatic Cervical Spinal Cord Injury Enrolled in the RISCIS Phase III Randomized Controlled Trial. J Neurotrauma. 2023 Sep;40(17-18):1889-1906. doi: 10.1089/neu.2022.0499. PMID 37130044
- [Derived] Nagoshi N, Nakashima H, Fehlings MG. Riluzole as a neuroprotective drug for spinal cord injury: from bench to bedside. Molecules. 2015 Apr 29;20(5):7775-89. doi: 10.3390/molecules20057775. PMID 25939067
- [Derived] Fehlings MG, Wilson JR, Frankowski RF, Toups EG, Aarabi B, Harrop JS, Shaffrey CI, Harkema SJ, Guest JD, Tator CH, Burau KD, Johnson MW, Grossman RG. Riluzole for the treatment of acute traumatic spinal cord injury: rationale for and design of the NACTN Phase I clinical trial. J Neurosurg Spine. 2012 Sep;17(1 Suppl):151-6. doi: 10.3171/2012.4.AOSPINE1259. PMID 22985381
- [Derived] Chow DS, Teng Y, Toups EG, Aarabi B, Harrop JS, Shaffrey CI, Johnson MM, Boakye M, Frankowski RF, Fehlings MG, Grossman RG. Pharmacology of riluzole in acute spinal cord injury. J Neurosurg Spine. 2012 Sep;17(1 Suppl):129-40. doi: 10.3171/2012.5.AOSPINE12112. PMID 22985379
- See also: The Reeve Foundation is dedicated to curing spinal cord injury by funding innovative research, and improving the quality of life for people living with paralysis through grants, information and advocacy. Click here for more information about the network. — http://christopherreeve.org